CLINICAL TRIAL: NCT00125255
Title: A Randomized, Double-blind, Placebo Controlled, Parallel Study Evaluating the Efficacy of S-Caine™ Peel (Lidocaine 7% and Tetracaine 7% Cream) for Induction of Local Dermal Anesthesia Before Vascular Access Procedures in Children
Brief Title: S-Caine™ Peel (Skin Numbing Cream) to Treat Pain During Vascular Access Procedures in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCP-46-05
Record Dates: First submitted 2005-07-27; First posted 2005-07-29 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- S-Caine Peel (Experimental)
  Interventions: Drug: S-Caine™ Peel (lidocaine and tetracaine cream 7%/7%)
- Placebo Peel (Placebo Comparator)
  Interventions: Drug: Placebo Peel

INTERVENTIONS:
Drug: S-Caine™ Peel (lidocaine and tetracaine cream 7%/7%) — S-Caine Peel comprising of a 1:1 eutectic mixture of 7% lidocaine and 7% tetracaine was applied topically. The study drug was applied at approximately 1 mm in thickness and remained on the treatment area for 30 minutes
  Other Names: Pliaglis
  Arms: S-Caine Peel
Drug: Placebo Peel — Placebo Peel applied topically at approximately 1 mm in thickness and remained on the treatment area for 30 minutes
  Other Names: Placebo
  Arms: Placebo Peel

SUMMARY:
The pain associated with medical procedures is often under-treated in children. Children often undergo painful procedures with little or no anesthetic, even when effective therapy is available. Reasons for not providing available therapy in children include concerns over adverse side effects as well as the length of time necessary to provide adequate anesthesia. Recent guidelines strongly advocate for the proactive treatment of pain in children, including the pain associated with medical procedures.

S-Caine™ Peel (lidocaine 7% and tetracaine 7% cream) is a eutectic formulation of lidocaine and tetracaine. The purpose of this study is to evaluate whether S-Caine Peel is effective in providing topical local dermal anesthesia prior to a vascular access procedure in children 5 through 17 years of age.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled, parallel study that evaluated the effectiveness of S-Caine Peel in providing local dermal anesthesia for vascular access procedures in children who were 5 through 17 years of age. Patients were randomized 1:1 to receive either one application of S-Caine Peel or one application of placebo for 30 minutes prior to a vascular access procedure.

During the screening visit, the study was fully explained to each patient's legal guardian and written informed consent was obtained. Whenever possible, patients provided assent. The screening visit also included: evaluating eligibility criteria; obtaining a medical history (including skin type, demographic data, and concomitant medications); obtaining a brief physical examination and urine pregnancy test (for females of childbearing potential), which had to be negative for the patient to enroll in the study; and providing patient education on how to assess pain using the Colored Analog Scale (CAS). The screening visit could occur on the same day as the procedure visit.

Upon meeting the eligibility criteria and completing the screening visit, patients were assigned the next available sequential patient number in their age group (5-11 years or 12-17 years). Based upon a randomized code, patients were randomized to receive either S Caine Peel or placebo for 30 minutes before the scheduled vascular access procedure.

The study drug application site could be on either the patient's left or right antecubital surface and covered an area of 10 cm2. A thin layer (approximately 1 mm or the thickness of a dime) of the study drug was applied evenly across the area to be treated for 30 minutes. Immediately following removal of the study drug, the study drug application site was evaluated for erythema, edema, blanching or other skin reactions. The vascular access procedure was then performed.

Upon completion of the vascular access procedure, the investigator's evaluation of procedural pain intensity and assessment of the adequacy of the anesthesia provided by the study drug were completed. Following these assessments, patients assessed their procedural pain intensity using the CAS. All pain evaluations were completed after the first attempt to gain vascular access. If the first attempt was unsuccessful and further attempts were required, the procedure was stopped and all pain assessments were performed before further attempts at vascular access were made.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 5 through 17 years of age.
* Patient has a medical indication to undergo a venous vascular access procedure (excluding peripherally inserted central catheter [PICC] lines) on the antecubital surface.

Exclusion Criteria:

* Patient is pregnant or breastfeeding.
* Patient has participated in a clinical trial of an unapproved drug within the previous 30 days.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2005-06; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 30 minutes
  The primary efficacy variable was pain intensity as reported by the patient using the Colored Analog Scale (CAS) (scale 0 to 10), a validated tool for measuring pain in children.

SECONDARY OUTCOMES:
Number of participants with adverse events | 30 minutes
  To monitor the nature and frequency of adverse events (AEs) associated with the application of S-Caine Peel

CONTACTS AND LOCATIONS:
Overall Officials: Susan T. Verghese, MD, Principal Investigator — Children's National Research Institute; Navil Sethna, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Andrew Wiznia, MD, Principal Investigator — Jacobi Medical Center
Locations (1):
- Children's Hospital, Boston, Massachusetts, United States